CLINICAL TRIAL: NCT04473014
Title: Towards a Deeper Understanding of Chronic Pediatric Pain: Exploring the Role of Sensory Processing Sensitivity
Brief Title: The Role of Sensory Processing Sensitivity in Pediatric Chronic Pain
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Helen Koechlin, Adjunct Senior Researcher, University Hospital, Basel, Switzerland
Other Study IDs: Heat Pain
Record Dates: First submitted 2020-06-30; First posted 2020-07-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
Keywords: sensory processing sensitivity
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Positive Mood: This group will be exposed to a positive mood induction prior to heat pain.
  Interventions: Behavioral: Heat Pain Paradigm
- Negative Mood: This group will be exposed to a negative mood induction prior to heat pain.
  Interventions: Behavioral: Heat Pain Paradigm
- Neutral Mood: This group will be exposed to a neutral mood induction prior to heat pain.
  Interventions: Behavioral: Heat Pain Paradigm

INTERVENTIONS:
Behavioral: Heat Pain Paradigm — A standardized heat pain paradigm will be applied. Pain threshold will be determined with the self-controlled search method starting at 32°C, with a mouse-click-induced increase of 0.1°C per click. Pain tolerance is defined as the time in seconds elapsed from the onset of the pain stimulus to a participant's withdrawal from the stimulus. Participants will be instructed to continue with the task for as long as they can and to press a button if it becomes too uncomfortable or painful. Temperature will then return to baseline. To avoid physical injury, the measurement will stop automatically at a maximum temperature of 50°C.

SUMMARY:
The aim of this project is to increase scientific understanding of whether the trait of SPS can help explain increased pain sensitivity and hence vulnerability for chronic pain. Additionally, it will be tested whether participants with high SPS report differences in pain intensity in response to positive, negative, or neutral mood induction compared to individuals with lower SPS.

DETAILED DESCRIPTION:
Background: Pain is defined as an unpleasant sensory and emotional experience and in its chronic form, pain is highly prevalent, up to 25% of children and adolescents are affected by it. The exact etiology of many forms of chronic pain remains unknown. One mechanism that has been proposed to underlie increased pain sensitivity is central sensitization, i.e., increased efficacy of the nervous system in transmitting pain signals, which manifests itself as a lower pain threshold. A lower pain threshold in turn has been recognized as a risk factor for the development of chronic pain. Being more sensitive to pain is one feature commonly shared by those with high sensory processing sensitivity (SPS), who are thought to react more strongly to both positive and negative environmental influences. The relationship between this increased sensitivity and pain tolerance has not been studied to date, but could contribute to our understanding of why some children and adolescents are more vulnerable to developing chronic pain than others.

Objectives and Aims: The aim of this project is to increase scientific understanding of whether the trait of SPS can help explain increased pain sensitivity and hence vulnerability for chronic pain. Additionally, it will be tested whether participants with high SPS report differences in pain intensity in response to positive, negative, or neutral mood induction compared to individuals with lower SPS.

Methods: To examine differences in pain perception of an experimentally induced pain stimulus between people with varying levels of SPS and whether pain perception can modulated by positive, negative, or neutral mood induction, I will apply a heat pain paradigm in a sample of healthy adolescents. Participants will be randomized to either neutral, positive or negative mood induction and I will test whether their pain sensitivity differs as a function of their scores on a high sensitivity scale and with regard to mood induction.

Expected Results: We expect highly sensitive adolescents to have a lower pain threshold and tolerance and to react more strongly to positive (with decreased pain ratings) and negative (with increased pain ratings) mood induction compared to those with lower scores on the sensitivity scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents aged 16-19 years

Exclusion Criteria:

* Chronic pain or another chronic condition
* Skin pathologies
* Sensory abnormalities affecting the tactile or thermal modality
* Pregnancy
* Current medication
* Current psychological or psychiatric treatment
* Insufficient language skills to understand the instructions

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited from local schools and at the University of Basel, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Pain Threshold | 1 day
  Temperature point where participants feel it changing from "hot" to "painful"
Pain Tolerance | 1 day
  the time in seconds elapsed from the onset of the pain stimulus to a participant's withdrawal from the stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Helen Koechlin, PhD, Principal Investigator — University of Basel, Switzerland; Boston Children's Hospital, Boston, MA, USA
Locations (1):
- Faculty of Psychology, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided